CLINICAL TRIAL: NCT02112240
Title: Novel Sentinel Lymph Node Mapping Technique in Early Stage Rectal Cancer
Brief Title: Feasibility Study to Develop Sentinel Lymph Node Mapping in Rectal Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No accrual. New study opening with modified technique.
Sponsor: University of Virginia (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Traci Hedrick, MD, Assistant Professor of Surgery, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16746
Record Dates: First submitted 2014-03-20; First posted 2014-04-11 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Rectal Cancer
Keywords: sentinel lymph node; lymphatic mapping; rectal tumor
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgery with pre- and intra-op imaging (Experimental): Subjects will have a preoperative flexible sigmoidoscopy where they will receive an endoscopic injection of 99mTc-sulfur colloid (up to 0.5 mCi) and 3 to 5 cc of circumferential endoscopic injections of Spot. A SPECT/CT will be performed prior to surgery to identify lymph nodes in the rectum. Subjects will proceed to their standard surgery. Intraoperative mobile gamma camera imaging of the rectum will occur before and after resection in attempt to identify sentinel lymph nodes.
  Interventions: Other: Intraoperative Mobile Gamma Camera imaging; Drug: Endoscopic injection of 99mTc-sulfur colloid; Other: Endoscopic injections of Spot; Procedure: Preoperative flexible sigmoidoscopy; Radiation: SPECT/CT

INTERVENTIONS:
Other: Intraoperative Mobile Gamma Camera imaging — Intraoperative images will be taken with a unique mobile gamma camera to identify sentinel lymph nodes in the rectum.
Drug: Endoscopic injection of 99mTc-sulfur colloid — Radiotracer injection around the rectal tumor for pre- and intra-operative imaging.
  Other Names: Tc-sulfur colloid
Other: Endoscopic injections of Spot — Dye injection for tattooing rectal tumor prior to surgical resection.
Procedure: Preoperative flexible sigmoidoscopy — Flexible sigmoidoscopy prior to surgery to facilitate endoscopic injections of radiotracer and dye.
Radiation: SPECT/CT — Preoperative imaging to identify lymph nodes in rectum.

SUMMARY:
The purpose of this study is to see if investigators can develop a technique to identify sentinel lymph nodes in the rectum for rectal cancer patients with the use of a radiotracer (Tc-sulfur colloid), a dye (Spot), and imaging, both pre- and intraoperatively. Eligible patients are those with stage I-III rectal cancer undergoing standard low anterior resection or abdominoperineal resection.

Investigators hypothesize that use of a unique intraoperative lymphatic mapping technique using a mobile gamma camera will identify the sentinel lymph node in patients with rectal cancer with greater than 80% sensitivity.

Subjects will receive injections of the tracer and dye prior to surgery, have preoperative SPECT/CT imaging to be used as a guide to the rectal lymphatic system and then proceed to their scheduled surgery. During surgery, images of the rectum will be taken with a unique mobile gamma camera prior to removal and upon resection.

If surgeons are able to identify the sentinel lymph nodes surrounding the rectal tumor, the hope is to combine this technique with a less invasive surgery called transanal endoscopic microsurgery (TEM) for early stage rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with stage I,II, or III rectal cancer undergoing standard trans- abdominal low anterior resection or abdominoperineal resection surgery at the University of Virginia
* Willing and able to give written informed consent

Exclusion Criteria:

* Patients less than 18 years of age
* Women who are pregnant and/or breastfeeding
* Prisoners
* Unable to give written informed consent
* Participants with medical contradictions or have potential problems complying with the requirements of the protocol, in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Evaluating the sensitivity of identifying the sentinel lymph node using a unique mobile gamma camera intraoperatively. | At the time of surgery and the time of pathological review, an expected average of 7 days.
  The primary endpoint is the sensitivity of sentinel lymph node (SLN) detection by the technique which will be estimated by the number of SLNs detected by the technique divided by the number noted at surgery or on final pathology review. 90% confidences interval around the estimate will help guide interpretation of the results.

SECONDARY OUTCOMES:
Feasibility | From the time of tracer and dye injections to 30 day postoperative visit
  Descriptive summaries will be used to list any complications that may have occurred pre-, intra- or post-operatively. Frequency and location of the sentinel lymph node (SLN) with respect to the tumor prior to surgery will be noted. In addition the location of the SLN in relation to the tumor will be documented during pathologic examination with the pathologist and surgeon to assess the feasibility of excision with transanal endoscopic microsurgery.

CONTACTS AND LOCATIONS:
Overall Officials: Traci L Hedrick, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States